CLINICAL TRIAL: NCT05862740
Title: ULTRA-LAP Trial: Laparoscopic Debulking Surgery (LDS) in Advanced Ovarian Cancer: a Feasibility Prospective Study
Brief Title: ULTRA-LAP Trial: Laparoscopic Debulking Surgery (LDS) in Advanced Ovarian Cancer
Acronym: ULTRA-LAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Roberto Tozzi, Professor and Chair, Azienda Ospedaliera di Padova
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 5497/AO/22; AOP2674 (Other: University of Padova)
Record Dates: First submitted 2023-03-10; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Advanced ovarian cancer; Debulking surgery; Multivisceral surgery; Laparoscopic debulking surgery
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Group A is the study group (completed laparoscopic debulking); Group B (conversion to laparotomy) is the control group in which laparoscopy could not be completed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic debulking surgery - LDS (Experimental): Primary debulking surgery or Interval debulking surgery performed by laparoscopy (P-LDS and I-LDS)
  Interventions: Procedure: Laparoscopic Debulking Surgery in advanced ovarian cancer
- Debulking surgery - DS (Active Comparator): Primary debulking surgery or Interval debulking surgery performed by/converted to laparotomy (PDS and IDS)
  Interventions: Procedure: Standard laparotomic Debulking Surgery in advanced ovarian cancer

INTERVENTIONS:
Procedure: Laparoscopic Debulking Surgery in advanced ovarian cancer — Laparoscopic debulking will be conducted until the surgical target is achieved or the operation is converted to laparotomy.
  Arms: Laparoscopic debulking surgery - LDS
Procedure: Standard laparotomic Debulking Surgery in advanced ovarian cancer — Debulking by laparotomy in patients when debulking could not be accomplished by laparoscopy.
  Arms: Debulking surgery - DS

SUMMARY:
ULTRA-LAP is a prospective study is to investigate the safety, efficacy and feasibility of laparoscopic debulking surgery (LDS) for the treatment of patients with advanced ovarian cancer.

The outcomes to measure are:

* Safety: the rate of patients experiencing intra- and post-operative early and late morbidities (within the hospitalization and up to 60 days from surgery)
* Efficacy: the rate of patients in which the surgical target set pre-operatively (complete resection) is achieved by laparoscopy.
* Feasibility: the rate of patients who have their procedure completed by laparoscopy

Patients will undergo laparoscopic debulking surgery (LDS) if the surgical target can be met. If it cannot be achieved by laparoscopy the surgeon will convert to laparotomy.

DETAILED DESCRIPTION:
The investigators intend to perform a prospective feasibility study on patients with primary diagnosis of advanced ovarian cancer (stage II to IV according to FIGO classification) who are referred to the tertiary cancer centre of the study. The latter is the Department of Gynecology and Obstetrics - Division of Women's and Children's Health - University of Padova - Italy. The statistical sample size calculation identified a minimum of 62 patients. The anticipated enrollment period will be about 4 years.

To confirm the ultimate eligibility to surgery and recruitment in the study, all patients undergo an exploratory laparoscopy (EXL).

The ideal surgical target is complete resection (CR) of all visible disease. Patients who are deemed not amenable to a CR at EXL will start neo-adjuvant chemotherapy. They will be reconsidered for the ULTRA-LAP study at time of interval surgery after 3 cycles of chemotherapy. Criteria for eligibility after neo-adjuvant chemotherapy are the same as per up-front surgery.

All patients recruited in the ULTRA-LAP trial will be discussed at Gynaecologic Oncology Multidisciplinary team (MDT) meeting, where imaging is reviewed and management is agreed. Following MDT decision:

* A Gynaecologic Oncologist will discuss the standard management and the ULTRA-LAP trial at time of out-patient clinic
* The ULTRA-LAP leaflet and consent form will be provided to the patient together with an accurate explanation of the study
* If the patient accepts to enter the study, a study registration form will be filled
* Participation in the study will be confirmed and the forms signed at time of pre-operative assessment and again confirmed at time of in-patient admission ULTRA-LAP trail will include all surgical procedures necessary to accomplish a complete resection (CR) of disease. The most common procedures necessary to obtain a CR are defined by The European Society of Gynaecological Oncology (ESGO), Society of Gynecologic Oncology (SGO) and the The National Institute for Health and Care Excellence (NICE) guidelines. All procedures will be performed by an expert Gynaecologic Oncologist with proven experience and high skills levels in oncological surgery. Once the surgeon realizes that a CR could not be achieved by laparoscopy, but prove to be feasible by laparotomy, the surgery is immediately converted to laparotomy.

Subsequent follow-up:

1. During Recovery:

   - The patients are going to be monitored daily and any relevant complications will be registered, graded (according to Clavien-Dindo classification) and treated.
2. Post recovery:

   * 1 st follow-up visit: At time of hospital's discharge an examination will be performed and, if necessary, further exams will be prescribed as appropriate.
   * 2 nd follow-up visit: following discharge, the next appointment is in the outpatient clinic roughly 15-20 days from the surgery.
   * 3 rd and last visit: at 30 days from the surgery a further appointment will be carried.

At each follow-up appointment the following will be registered:

* Occurrence of complications
* Physical examination
* Changes in normal quality of life.

Achievement of a CR will be determined at time of surgery and confirmed by a pre-chemotherapy CT scan. Should discrepancy arise, CT scan will be reviewed at MDT.

All patients will be closely monitored with a rigorous follow-up program every 90 days for the first two years and then every 120 days for the subsequent 2 years. In addition, all patient could contact the department if any unexpected complications happens between follow-up time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced epithelial ovarian cancer (II-IV Stage FIGO) candidates to PDS (primary debulking surgery) or IDS (interval debulking surgery: neoadjuvant chemotherapy followed by IDS).
* Participant is willing and able to give informed consent for participation in the study.
* Female aged 18 years or above.
* Primary diagnosis of advanced epithelial ovarian cancer (tubal and peritoneal cancer included).

Exclusion Criteria:

* Comorbidities non-allowing for radical surgery
* Poor Performance Status (Karnofsky Index < 70)
* Concomitant or past history of malignancy, regardless of treatment status
* Recent or past story of pancreatitis or hepatitis
* Recent or past story of pleural effusion or lung injuries or respiratory failure
* Cardiac major pathologies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety: rate of complications/morbidities | 60 days
  Safety will be measured as the rate of patients experiencing intra- and post-operative early and late morbidities (within and after the hospitalization up to 60 days from surgery) and it will be compared to the morbidity rate of patients having similar surgery by laparotomy. Complications are going to be graded according to Clavien-Dindo classification.
Efficacy: rate of complete resection (CR) in group 1 | 60 days
  Efficacy will be measured as the rate of patients in which the surgical target set pre-operatively is achieved by laparoscopy.
Feasibility: rate of procedures completed by laparoscopy | 60 days
  Feasibility will be measured as the rate of patients who have their procedure completed by laparoscopy.

SECONDARY OUTCOMES:
Progression Free Survival (PFS). | 5 years
  the time interval from the surgical treatment to the date of the documented first recurrence of disease, by CA 125 (Carbohydrate Antigen 125) and/or CT scan.
Overall Survival (OS). | 5 years
  time between surgery and death.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Tozzi, Professor, Principal Investigator — Azienda Ospedale Università di Padova
Locations (1):
- Azienda Ospedaliera Universitaria di Padova,, Padua, Padova, Veneto, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elattar A, Bryant A, Winter-Roach BA, Hatem M, Naik R. Optimal primary surgical treatment for advanced epithelial ovarian cancer. Cochrane Database Syst Rev. 2011 Aug 10;2011(8):CD007565. doi: 10.1002/14651858.CD007565.pub2. PMID 21833960
- [Result] Shih KK, Chi DS. Maximal cytoreductive effort in epithelial ovarian cancer surgery. J Gynecol Oncol. 2010 Jun;21(2):75-80. doi: 10.3802/jgo.2010.21.2.75. Epub 2010 Jun 30. PMID 20613895
- [Result] Elstrand MB, Sandstad B, Oksefjell H, Davidson B, Trope CG. Prognostic significance of residual tumor in patients with epithelial ovarian carcinoma stage IV in a 20 year perspective. Acta Obstet Gynecol Scand. 2012 Mar;91(3):308-17. doi: 10.1111/j.1600-0412.2011.01316.x. Epub 2012 Jan 9. PMID 22050605
- [Result] Pomel C, Akladios C, Lambaudie E, Rouzier R, Ferron G, Lecuru F, Classe JM, Fourchotte V, Paillocher N, Wattiez A, Montoriol PF, Thivat E, Beguinot M, Canis M. Laparoscopic management of advanced epithelial ovarian cancer after neoadjuvant chemotherapy: a phase II prospective multicenter non-randomized trial (the CILOVE study). Int J Gynecol Cancer. 2021 Dec;31(12):1572-1578. doi: 10.1136/ijgc-2021-002888. Epub 2021 Oct 20. PMID 34670829
- [Result] Fagotti A, Gueli Alletti S, Corrado G, Cola E, Vizza E, Vieira M, Andrade CE, Tsunoda A, Favero G, Zapardiel I, Pasciuto T, Scambia G. The INTERNATIONAL MISSION study: minimally invasive surgery in ovarian neoplasms after neoadjuvant chemotherapy. Int J Gynecol Cancer. 2019 Jan;29(1):5-9. doi: 10.1136/ijgc-2018-000012. PMID 30640676
- [Derived] Tozzi R, Noventa M, Saccardi C, Spagnol G, De Tommasi O, Coldebella D, Marchetti M. Feasibility of laparoscopic Visceral-Peritoneal Debulking (L-VPD) in patients with stage III-IV ovarian cancer: the ULTRA-LAP trial pilot study. J Gynecol Oncol. 2024 Mar;35(2):e14. doi: 10.3802/jgo.2024.35.e14. Epub 2023 Oct 16. PMID 37921599